CLINICAL TRIAL: NCT01484366
Title: Prospective Randomized Trial for Forearm Shaft Fractures: Plating of Radius and Ulna vs. Plating of Radius and Nailing of Ulna
Brief Title: Forearm Shaft Fractures: Plating of Radius and Ulna Versus Plating of Radius and Nailing of Ulna
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment. Treament no longer used by researchers.
Sponsor: Florida Orthopaedic Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBFA
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Fractures of Radius and Ulna
Keywords: fractures of both radius and ulna
MeSH Terms: interventions — Fracture Fixation, Intramedullary; Electroplating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intramedullary nailing and plating (Active Comparator): intramedullary nailing of the ulna and plating of the radius in the treatment of both bone forearm fractures
  Interventions: Procedure: intramedullary nailing and plating
- plating (Active Comparator): plating of both the radius and ulna in the treatment of both bone forearm fractures
  Interventions: Procedure: plating

INTERVENTIONS:
Procedure: intramedullary nailing and plating — Surgical intramedullary nailing of the ulna and plating of the radius
  Other Names: forearm fractures
  Arms: intramedullary nailing and plating
Procedure: plating — Surgical plating of both bonforearm fractures
  Other Names: Forearm fractures
  Arms: plating

SUMMARY:
The hypothesis is that intramedullary nailing of the ulna and plating of the radius will result in a superior outcome as evidenced by two primary end points:

1. a lower rate of implant pain
2. a lower re-operation rate to remove painful hardware.

DETAILED DESCRIPTION:
This is a prospective, randomized study to determine if intramedullary nailing of the ulna and plating of the radius is equal to, or superior to plating of both the radius and ulna for the treatment of both bone forearm fractures.

ELIGIBILITY:
Inclusion Criteria:

* Diaphyseal fractures of both radius and ulna
* Ulna fractures that are oblique or transverse
* Fractures may be closed or Grade I-IIIA open
* Patients must be over 18 and skeletally mature

Exclusion Criteria:

* Children under the age of 18
* Pregnancy
* Comminuted ulna fractures
* Those with associated bony elbow or wrist trauma
* Elbow dislocation
* Subjects with bone pathology (osteoporosis, OI, Paget's disease, bone cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
implant pain | 1 year
  a visual analog scale (VAS) will be used to assess pain in the forearm

SECONDARY OUTCOMES:
re-operation rate to remove painful hardware | 1 year
  repeat surgical intervention will be captured

CONTACTS AND LOCATIONS:
Overall Officials: Roy Sanders, MD, Principal Investigator — Florida Orthopaedic Institute
Locations (2):
- United States (2):
  - Tampa General Hospital, Tampa, Florida
  - St Josephs Hospital, Tampa, Florida